CLINICAL TRIAL: NCT04731428
Title: The Effect of Progressive Relaxation Exercise on Physiological Parameters, Pain and Anxiety in Patients Undergoing Colorectal Cancer Surgery: A Randomized Controlled Study
Brief Title: Effect of Progressive Relaxation Exercise on Physiological Parameters, Pain, Anxiety in Colorectal Cancer Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: YASEMİN ÖZHANLI (Other)
Responsible Party: Sponsor-Investigator, YASEMİN ÖZHANLI, Research Assistant Doctor, Kocaeli University
Organization: Kocaeli University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 2018/141525
Record Dates: First submitted 2021-01-15; First posted 2021-02-01 (Actual); Last update posted 2021-02-01 (Actual); Status verified 2021-01

CONDITIONS: Postoperative Pain; Nursing Caries; Anxiety
Keywords: Progressive relaxation exercise; Colorectal cancer surgery; Pain; Anxiety; Nursing care
MeSH Terms: conditions — Pain, Postoperative; Anxiety Disorders; Pain

STUDY DESIGN:
Intervention Model Description: Randomized Controlled Study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Progressive Relaxation Exercise (Experimental): In individuals with normal daily circadian rhythms, cortisol levels peak at 8:00 AM, followed by a constantly declining daily cycle throughout the day. Therefore, it is important to collect blood samples taken for the measurement of serum cortisol levels approximately at the same time. Venous blood samples (3 ml) were obtained from the upper arm at 06:45 AM to evaluate the baseline and 45 minutes after Progressive Relaxation Exercise at 08:00. Vital signs and oxygen saturation were assessed at 6:30 AM before Progressive Relaxation Exercise and at 07:20 AM 5 minutes after Progressive Relaxation Exercise. Measurements were performed in the morning on the day of surgery and on postoperative days 1, 2, and 3.
  Interventions: Behavioral: Progressive Relaxation Exercise
- Standard Care (No Intervention): In the control group, no application made during and after the surgical intervention, and routine treatment and care applied.

INTERVENTIONS:
Behavioral: Progressive Relaxation Exercise — Progressive Relaxation Exercise involves stretching sixteen muscle groups while breathing in sequentially, relaxing while exhaling. Exercise can be from head to toe or from foot to head. In order for the technique to be effective, it is important to have affective (music, etc.) and visual aids. During the exercise, the patient should complete the processes of perceiving the tension in his body, maintaining control and getting into a state of relaxation. After the patient is informed about the exercise, the person starts with breathing exercises. A deep but relaxing breath is taken from the nose, and lips are given by contracting simultaneously with relaxation. During this application, the patient keeps contracting the muscle group that he exercises for 10 seconds; the nurse provides the patient to notice the temperature / warming felt in the muscle group.
  Arms: Progressive Relaxation Exercise

SUMMARY:
This research was carried out as an pre-test/post-test control group experimental design study in order to determine the effect of progressive relaxation exercises on the level of vital sign, pain and anxiety underwent who laparoscopic surgery for colorectal cancer in patients. This research data was collected between March 2018 and May 2019. The research was carried out with 63 patients (experiment group= 31, control group= 32) who underwent elective laparoscopic colorectal surgery in a general surgery clinic of a university hospital in Istanbul and in accordance with the research criteria. Patients in the experiment group were taught breathing exercises in the preoperative period and on the 1st, 2nd and 3rd day after surgery then, progressive relaxation exercise that lasted 15 minutes was applied to the group. Pain (Short McGill Pain Scale) and anxiety (STAI-S Scale) levels of both groups were evaluated in the preoperative and postoperative period. The patient's vital signs, oxygen saturation and serum cortisol level parameters were measured in the same time interval before and after the relaxation exercise. Significance was evaluated at p <0.05 and p<0,001 levels in the analysis of the data. Prior to the study, the consent of the institution and ethics committee, written and verbal patient consent were obtained.

DETAILED DESCRIPTION:
The universe of the study consisted of patients with colorectal cancer who were admitted to Istanbul University, Istanbul Faculty of Medicine, General Surgery Clinics for treatment between March 2018 and May 2019 and who would undergo laparoscopic surgery.The research was planned as a randomized controlled experimental study. Block randomization method was to determine the experimental and control groups. In order for the groups to be distributed homogeneously, the order produced by a computer program(https://www.randomizer.org/) was used. Randomization done by a biostatistician outside the researcher. Patients who meet the inclusion criteria and agree to participate in the study assigned to the experimental and control groups according the randomization list.Research data will be collected in a hospital's general surgery ward between March 2018 and May 2019. The independent variable of the study is Progressive Relaxation Exercise.The dependent variables of the study are physiological parameters, pain, anxiety and serum cortisol. In the research, "Individual Characteristics Form" and "Patient Follow-up Form" prepared by the researcher in line with the literature will be used as data collection tools.

ELIGIBILITY:
Inclusion Criteria:

* Being 18 years or over,
* Consenting to participate in the study with verbal and written declaration after being informed,
* Being scheduled for elective laparoscopic colorectal cancer surgery,
* Not participating in another randomized controlled study simultaneously.

Exclusion Criteria:

* Having a health problem that will alter cortisol release,
* Preoperative and postoperative unconsciousness,
* Having a psychiatric problem,
* Having a disease that requires corticosteroid therapy,
* Developing any complications during the operation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 63 (Actual)
Dates: Start 2018-03-15 (Actual); Primary Completion 2019-05-30 (Actual); Study Completion 2020-06-10 (Actual)

PRIMARY OUTCOMES:
Preoperative pain severity | Preoperative pain assessment of the groups was made 2 hours before surgery.
  Pain severity assessment with Short Form McGill Pain Questionnaire In the first part, pain intensity is evaluated as 0=no pain, 1=mild pain, 2=moderate pain, 3=severe pain In the second part, the pain felt is evalauted using the Visuel Analog Scale (VAS).0-10; 0- No Pain, 10- Worst pain In the third part, the total pain intensity is measured with a 6-point Likert-type assessment. (0=no pain, 1=mild, 2=annoying , 3=troublesome, 4=miserable, 5=unbearable pain) Pain assessment for the experimental group Preoperative pain assessment of the experimental group was made before applying the progressive relaxation exercise. This evaluation was made 2 hours before surgery (6.30 am).
  Pain assessment for the control group Preoperative pain assessment of the control group was made 2 hours before the operation in order to ensure the equivalence between the groups (6.30 am).
Preoperative anxiety severity | Preoperative anxiety assessment of the groups was made 2 hours before surgery.
  Anxiety severity with Spielberger's State and Trait Anxiety Inventory State Anxiety Subscale are specified by choosing one of the options "1) not at all, 2) somewhat, 3) moderately so, and 4) very much so" according to the severity of such experiences.
  Anxiety assessment for the experimental group Preoperative anxiety assessment of the experimental group was made before applying the progressive relaxation exercise. This evaluation was made 2 hours before surgery (6.30 am).
  Anxiety assessment for the control group Preoperative anxiety assessment of the control group was made 2 hours before the operation in order to ensure the equivalence between the groups (6.30 am).
Preoperative systolic and diastolic blood pressure (mmHg) (1st. assessment) | In the preoperative period, systolic and diastolic blood pressure (mmHg) evaluations were made 2 hours before surgery.
  Systolic and diastolic blood pressure (mmHg) evaluations were made with a digital blood pressure measuring device.
  For experimental group The first evaluation was made before applying the progressive relaxation exercise(6.30 am).
  For the control group The first evaluation was made 6.30am.
Preoperative pulse rate (heart rate per minute) (1st. assessment) | In the preoperative period, the pulse rate was evaluated 2 hours before surgery.
  Pulse rate (heart rate per minute) evaluation was made with a digital pulse-meter.
  For the experimental group The first evaluation was made before applying the progressive relaxation exercise (6.30 am).
  For the control group The first evaluation was made 6.30am.
Preoperative respiratory rate (respiratory per minute) (1st. assessment) | In the preoperative period, respiratory rate was evaluated 2 hours before surgery.
  Respiratory rate (respiratory per minute) evaluation was made by the researcher by counting 1 minute.
  For the experimental group The first evaluation was made before applying the progressive relaxation exercise (6.30am).
  For the control group The first evaluation was made 6.30am.
Preoperative body temperature (Celcius) (1st. assessment) | In the preoperative period, body temperature was evaluated 2 hours before surgery
  Body temperature (Celcius)assessment was made with a digital thermometer. For the experimental group The first evaluation was made before applying the progressive relaxation exercise (6.30am).
  For the control group The first evaluation was made 6.30am.
Preoperative oxygen saturation (SpO2) (1st. assessment) | In the preoperative period, oxygen saturation was evaluated 2 hours before surgery.
  Oxygen saturation (SpO2) was evaluated with a pulse oximeter. For the experimental group The first evaluation was made before applying the progressive relaxation exercise (6.30am).
  For the control group The first evaluation was made 6.30am.
Preoperative serum cortisol levels (1st. assessment) | In the preoperative period, serum cortisol levels assessment of the groups was made 2 hours before surgery.
  Blood samples were placed in tubes containing separator gel (SST-yellow tube) and serum cortisol level was analyzed in the relevant laboratory.
  For the experimental group The first evaluation was made before applying the progressive relaxation exercise (6.45 am).
  For the control group The first evaluation was made 6.45am.
Use of analgesic (See Table 1)(in the first 24 hours after surgery) | Analgesic consumption of the patients was recorded in the first 24 hours after surgery.
  In this section, dose (mg) of use of analgesics were followed. Table 1: Monitoring of analgesic use of patients Analgesic name Dose (mg) Postoperative 0 Opioid NSAİ Other
Preoperative systolic and diastolic blood pressure (mmHg) (2nd. assessment) | In the preoperative period, systolic and diastolic blood pressure (mmHg) evaluations were made 1 hour before surgery.
  Systolic and diastolic blood pressure (mmHg) evaluations were made with a digital blood pressure measuring device.
  For experimental group Progressive relaxation exercise was applied, the second evaluation was made 5 minutes after the application (7.20am.).
  For the control group Progressive relaxation exercise wasn't applied because of was control group, the second evaluation was made 7.20am.
Preoperative pulse rate (heart rate per minute) (2nd. assessment) | In the preoperative period, the pulse rate was evaluated 1 hour before surgery.
  Respiratory rate (respiratory per minute) evaluation was made by the researcher by counting 1 minute.
  For the experimental group Progressive relaxation exercise was applied, the second evaluation was made 5 minutes after the application (7.20am.).
  For the control group Progressive relaxation exercise wasn't applied because of was control group, the second evaluation was made 7.20am.
Preoperative respiratory rate (respiratory per minute) (2nd. assessment) | In the preoperative period, respiratory rate was evaluated 1 hour before surgery.
  Respiratory rate (respiratory per minute) evaluation was made by the researcher by counting 1 minute.
  For the experimental group Progressive relaxation exercise was applied, the second evaluation was made 5 minutes after the application (7.20am.).
  For the control group Progressive relaxation exercise wasn't applied because of was control group, the second evaluation was made 7.20am.
Preoperative body temperature (Celcius) (2nd. assessment) | In the preoperative period, body temperature was evaluated 1 hour before surgery.
  Body temperature (Celcius)assessment was made with a digital thermometer. For the experimental group Progressive relaxation exercise was applied, the second evaluation was made 5 minutes after the application (7.20am.).
  For the control group Progressive relaxation exercise wasn't applied because of was control group, the second evaluation was made 7.20am.
Preoperative oxygen saturation (SpO2) (2nd. assessment) | In the preoperative period, oxygen saturation was evaluated 1 hour before surgery.
  Oxygen saturation (SpO2) was evaluated with a pulse oximeter. For the experimental group Progressive relaxation exercise was applied, the second evaluation was made 5 minutes after the application (7.20am.).
  For the control group Progressive relaxation exercise wasn't applied because of was control group, the second evaluation was made 7.20am.
Preoperative serum cortisol levels (2nd. assessment) | In the preoperative period, serum cortisol levels assessment of the groups was made 1 hour before surgery.
  Blood samples were placed in tubes containing separator gel (SST-yellow tube) and serum cortisol level was analyzed in the relevant laboratory.
  For the experimental group Progressive relaxation exercise was applied, the second evaluation was made 45 minutes after the application (8.00am.).
  For the control group Progressive relaxation exercise wasn't applied because of was control group, the second evaluation was made 8.00am.
Use of analgesic (See Table 1)(postoperative 1st. day) | Analgesic consumption of the patients was recorded in the postoperative 1st. day.
  In this section, dose of use of analgesics were followed. Table 1: Monitoring of analgesic use of patients Analgesic name Doses (mg) Postoperative 1 Opioid NSAİ Other
Use of analgesic (See Table 1)(postoperative 2nd day) | Analgesic consumption of the patients was recorded in the postoperative 2nd. day.
  In this section, dose of use of analgesics were followed. Table 1: Monitoring of analgesic use of patients Analgesic name Dose (mg) Postoperative 2 Opioid NSAİ Other
Use of analgesic (See Table 1)(postoperative 3rd day) | Analgesic consumption of the patients was recorded in the postoperative 3rd. days.
  In this section, dose of use of analgesics were followed. Table 1: Monitoring of analgesic use of patients Analgesic name Dose (mg) Postoperative 3 Opioid NSAİ Other

SECONDARY OUTCOMES:
Postoperative pain severity | Postoperative pain assessment of the groups was made postoperative 3rd. day.
  Pain severity assessment with Short Form McGill Pain Questionnaire
  For the experimental group The pain assessment of the experimental group in the postoperative period was made on the 3rd day after surgery. This evaluation was made 1 hour after the progressive relaxation exercise on the 3rd postoperative day (8.30 am).
  For the control group Postoperative pain assessment of the control group was made on the 3rd day after surgery.
  Postoperative pain assessment of the control group was made on the 3rd day after surgery. Post-operative pain assessment of the control group was performed at the same time (8.30 am) to ensure intergroup equivalence.
Postoperative anxiety severity | Postoperative anxiety assessment of the groups was made postoperative 3rd. day.
  Anxiety severity with Spielberger's State and Trait Anxiety Inventory State Anxiety Subscale are specified by choosing one of the options "1) not at all, 2) somewhat, 3) moderately so, and 4) very much so" according to the severity of such experiences.
  Anxiety assessment for the experimental group The anxiety assessment of the experimental group in the postoperative period was made on the 3rd day after surgery. This evaluation was made 1 hour after the progressive relaxation exercise on the 3rd postoperative day (8.30 am).
  Anxiety assessment for the control group Postoperative anxiety assessment of the control group was made on the 3rd day after surgery.
  Postoperative anxiety assessment of the control group was made on the 3rd day after surgery. Post-operative anxiety assessment of the control group was performed at the same time (8.30 am) to ensure intergroup equivalence.
Postoperative systolic and diastolic blood pressure (mmHg) (1st. assessment) | Systolic and diastolic blood pressure (mmHg) evaluations were made on postoperative 1st. day.
  Systolic and diastolic blood pressure (mmHg) evaluations were made with a digital blood pressure measuring device.
  For the experimental group Measurements were made before and after progressive relaxation exercise. For the control group The measurements of the control group were made at the same time as the measurements of the experimental group to ensure intergroup equivalence.
Postoperative systolic and diastolic blood pressure (mmHg) (2nd. assessment) | Systolic and diastolic blood pressure (mmHg) evaluations were made on postoperative 2nd. day.
  Systolic and diastolic blood pressure (mmHg) evaluations were made with a digital blood pressure measuring device.
  For the experimental group Measurements were made before and after progressive relaxation exercise. For the control group The measurements of the control group were made at the same time as the measurements of the experimental group to ensure intergroup equivalence.
Postoperative systolic and diastolic blood pressure (mmHg) (3rd. assessment) | Systolic and diastolic blood pressure (mmHg) evaluations were made on postoperative 3rd. day.
  Systolic and diastolic blood pressure (mmHg) evaluations were made with a digital blood pressure measuring device.
  For the experimental group Measurements were made before and after progressive relaxation exercise. For the control group The measurements of the control group were made at the same time as the measurements of the experimental group to ensure intergroup equivalence.
Postoperative pulse rate (heart rate per minute) (1st. assessment) | Pulse rate (heart rate per minute) evaluation was made on postoperative 1st. day.
  Pulse rate (heart rate per minute) evaluation was made with a digital pulse-meter.
  For the experimental group Measurements were made before and after progressive relaxation exercise. For the control group The measurements of the control group were made at the same time as the measurements of the experimental group to ensure intergroup equivalence.
Postoperative pulse rate (heart rate per minute) (2nd. assessment) | Pulse rate (heart rate per minute) evaluation was made on postoperative 2nd. day.
  Pulse rate (heart rate per minute) evaluation was made with a digital pulse-meter.
  For the experimental group Measurements were made before and after progressive relaxation exercise. For the control group The measurements of the control group were made at the same time as the measurements of the experimental group to ensure intergroup equivalence.
Postoperative pulse rate (heart rate per minute) (3rd. assessment) | Pulse rate (heart rate per minute) evaluation was made on postoperative 3rd. day.
  Pulse rate (heart rate per minute) evaluation was made with a digital pulse-meter.
  For the experimental group Measurements were made before and after progressive relaxation exercise. For the control group The measurements of the control group were made at the same time as the measurements of the experimental group to ensure intergroup equivalence.
Postoperative respiratory rate (respiratory per minute) (1st. assessment) | Respiratory rate (respiratory per minute) evaluations was made on postoperative 1st. day.
  Respiratory rate (respiratory per minute) evaluation was made by the researcher by counting 1 minute.
  For the experimental group Measurements were made before and after progressive relaxation exercise. For the control group The measurements of the control group were made at the same time as the measurements of the experimental group to ensure intergroup equivalence.
Postoperative respiratory rate (respiratory per minute) (2nd. assessment) | Respiratory rate (respiratory per minute) evaluations was made on postoperative 2nd. day.
  Respiratory rate (respiratory per minute) evaluation was made by the researcher by counting 1 minute.
  For the experimental group Measurements were made before and after progressive relaxation exercise. For the control group The measurements of the control group were made at the same time as the measurements of the experimental group to ensure intergroup equivalence.
Postoperative respiratory rate (respiratory per minute) (3rd. assessment) | Respiratory rate (respiratory per minute) evaluations was made on postoperative 3rd. day.
  Respiratory rate (respiratory per minute) evaluation was made by the researcher by counting 1 minute.
  For the experimental group Measurements were made before and after progressive relaxation exercise. For the control group The measurements of the control group were made at the same time as the measurements of the experimental group to ensure intergroup equivalence.
Postoperative body temperature (celcius) (1st. assessment) | Body temperature (0C) evaluation was made on postoperative 1st. day.
  Body temperature (celcius)assessment was made with a digital thermometer. For the experimental group Measurements were made before and after progressive relaxation exercise. For the control group The measurements of the control group were made at the same time as the measurements of the experimental group to ensure intergroup equivalence.
Postoperative body temperature (celcius) (2nd. assessment) | Body temperature (0C) evaluation was made on postoperative 2nd. day.
  Body temperature (celcius)assessment was made with a digital thermometer. For the experimental group Measurements were made before and after progressive relaxation exercise. For the control group The measurements of the control group were made at the same time as the measurements of the experimental group to ensure intergroup equivalence.
Postoperative body temperature (celcius) (3rd. assessment) | Body temperature (0C) evaluation was made on postoperative 3rd. day.
  Body temperature (celcius)assessment was made with a digital thermometer. For the experimental group Measurements were made before and after progressive relaxation exercise. For the control group The measurements of the control group were made at the same time as the measurements of the experimental group to ensure intergroup equivalence.
Postoperative oxygen saturation (SpO2) (1st. assessment) | Oxygen saturation (SpO2) evaluation was made on postoperative 1st. day.
  Oxygen saturation (SpO2) was evaluated with a pulse oximeter. For the experimental group Measurements were made before and after progressive relaxation exercise. For the control group The measurements of the control group were made at the same time as the measurements of the experimental group to ensure intergroup equivalence.
Postoperative oxygen saturation (SpO2) (2nd. assessment) | Oxygen saturation (SpO2) evaluation was made on postoperative 2nd. day.
  Oxygen saturation (SpO2) was evaluated with a pulse oximeter. For the experimental group Measurements were made before and after progressive relaxation exercise. For the control group The measurements of the control group were made at the same time as the measurements of the experimental group to ensure intergroup equivalence.
Postoperative oxygen saturation (SpO2) (3rd. assessment) | Oxygen saturation (SpO2) evaluation was made on postoperative 3rd. day.
  Oxygen saturation (SpO2) was evaluated with a pulse oximeter. For the experimental group Measurements were made before and after progressive relaxation exercise. For the control group The measurements of the control group were made at the same time as the measurements of the experimental group to ensure intergroup equivalence.
Postoperative serum cortisol levels (1st. assessment) | In the postoperative period, serum cortisol levels assessment of the groups was made on postoperative 1st. day.
  Blood samples were placed in tubes containing separator gel (SST-yellow tube) and serum cortisol level was analyzed in the relevant laboratory.
  For the experimental group The first day evaluation was made 45 minutes after applying the progressive relaxation exercise (8.00 am).
  For the control group The first day evaluation was made 8.00 am. Progressive relaxation exercise wasn't applied because of was control group.
Postoperative serum cortisol levels (2nd. assessment) | In the postoperative period, serum cortisol levels assessment of the groups was made on postoperative 2nd. day.
  Blood samples were placed in tubes containing separator gel (SST-yellow tube) and serum cortisol level was analyzed in the relevant laboratory.
  For the experimental group The second day evaluation was made 45 minutes after applying the progressive relaxation exercise (8.00 am).
  For the control group The second day evaluation was made 8.00 am. Progressive relaxation exercise wasn't applied because of was control group.
Postoperative serum cortisol levels (3rd. assessment) | In the postoperative period, serum cortisol levels assessment of the groups was made on postoperative 3rd. day.
  Blood samples were placed in tubes containing separator gel (SST-yellow tube) and serum cortisol level was analyzed in the relevant laboratory.
  For the experimental group The third day evaluation was made 45 minutes after applying the progressive relaxation exercise (8.00 am).
  For the control group The third day evaluation was made 8.00 am. Progressive relaxation exercise wasn't applied because of was control group.

CONTACTS AND LOCATIONS:
Overall Officials: Nuray Akyüz, Assoc. Prof., Study Director — Istanbul University - Cerrahpasa; Yasemin Özhanlı, PhD, Study Chair — Istanbul University - Cerrahpasa
Locations (1):
- Istanbul University-Istanbul Medical Faculty Hospital, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Ozhanli Y, Akyuz N. The Effect of Progressive Relaxation Exercise on Physiological Parameters, Pain and Anxiety Levels of Patients Undergoing Colorectal Cancer Surgery: A Randomized Controlled Study. J Perianesth Nurs. 2022 Apr;37(2):238-246. doi: 10.1016/j.jopan.2021.08.008. Epub 2021 Dec 10. PMID 34903440